CLINICAL TRIAL: NCT00229554
Title: Assessing and Addressing Patient Colorectal Cancer Screening Barriers
Brief Title: Survey of ColoRectal Cancer Education and Environment Needs
Acronym: SCREEN
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: IIR 04-042
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2009-01

CONDITIONS: Colorectal Neoplasms; Mass Screening; Patient Compliance
Keywords: health surveys; questionnaires
MeSH Terms: conditions — Colorectal Neoplasms; Patient Compliance

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Male and female veterans age 50-75 who have had one or more primary care visits at a VA Medical facility in the past two years.

SUMMARY:
Despite strong evidence for the effectiveness and cost-effectiveness of a variety of colorectal cancer (CRC) screening methods for reducing CRC mortality, current CRC screening rates fall far below the levels needed to significantly impact CRC mortality. Unfortunately, however, the existing literature on patient CRC screening behavior does not yet provide a sufficient evidence base for making sound recommendations regarding how to most effectively improve upon these rates in the VA. This study will inform future CRC screening promotion efforts and make important scientific contributions to existing literature by: (a) delineating the relative contribution of patient cognitive, environmental and background factors to CRC screening behavior using a multi-level, theory driven analysis approach on a nationally representative sample, and (b) identifying the determinants of variation in CRC screening behavior across vulnerable population subgroups.

DETAILED DESCRIPTION:
Background / Rationale:

Despite strong evidence for the effectiveness and cost-effectiveness of a variety of colorectal cancer (CRC) screening methods for reducing CRC mortality, current CRC screening rates fall far below the levels needed to significantly impact CRC mortality. Unfortunately, however, the existing literature on patient CRC screening behavior does not yet provide a sufficient evidence base for making sound recommendations regarding how to most effectively improve upon these rates in the VA. This study will inform future CRC screening promotion efforts and make important scientific contributions to existing literature by: (a) delineating the relative contribution of patient cognitive, environmental and background factors to CRC screening behavior using a multi-level, theory driven analysis approach on a nationally representative sample, and (b) identifying the determinants of variation in CRC screening behavior across vulnerable population subgroups.

Objective(s):

The overall goal of this study was to address significant gaps in the existing evidence base in order to inform the development of effective patient-directed interventions to increase CRC screening among veterans age 50 and older. This was accomplished by using data collected from a mailed patient survey and theory-based analysis approaches to uncover key barriers to screening adherence and to identify fruitful intervention approaches for modifying them. The specific primary objectives of this study were to: (1) Estimate the relative effect of patient cognitive (knowledge, attitudes, and self-efficacy), environmental (social network and medical care characteristics), and background (demographics, health status, prior screening experiences) factors on CRC screening behavior; (2) Identify factors that contribute to any disparities in CRC screening behavior by race/ethnicity or other patient characteristics; (3) Identify from these analyses: (a) priority population subgroups to target in future interventions (i.e., those at the greatest risk of failing to be screened), and (b) priority factors to target in future interventions (i.e., those that are not only strongly associated with CRC screening but also prevalent in the target population and amenable to intervention, as well as those that are most likely to ameliorate race and other disparities). Secondary objectives included: (1) assessing patient values and preferences regarding the various CRC screening modality options, (2) estimating stage of readiness to adopt CRC screening in the study population, and (3) validating measures of CRC knowledge and self-reported screening behavior.

Methods:

This is an observational study based on a nationally representative, cross-sectional mailed survey of 3,744 male and female veterans age 50-75 who have had one or more primary care visits at a VA Medical facility in the past two years. The survey sample was drawn using a two stage procedure where we first randomly select 24 VA facilities stratified by size and racial mix and then select a simple random sample of 156 eligible veterans from each sampled facility. Prior to the national survey, a pilot survey was conducted with the purpose of refining both the study instruments and the study protocol. The sample consisted of 900 randomly selected veterans from the Minneapolis VA Medical Center meeting the same sampling eligibility criteria used for the national mailed survey. The mailed patient questionnaire, made up primarily of previously validated measures, included measures of self-reported CRC screening behavior; patient demographic, health, social network and medical care characteristics; CRC screening knowledge, attitudes, social norms and self-efficacy; and attitudes toward medical care. Additional measures of organizational-level CRC screening practices from a recently completed VA facility survey were linked to the patient survey.The primary outcome is whether the patient is currently compliant with CRC screening guidelines (i.e., received either a fecal occult blood test in the past year, a sigmoidoscopy or double contrast barium enema in the past five years, or a colonoscopy in the past ten years). The primary analyses tested (using logistic regression and a multi-level, structural equation modeling approach) specific hypotheses about the association between this measure and patient background, cognitive and environmental factors and their interactions. Additional analyses conducted include a multinomial logistic regression to assess patient screening mode preferences and their determinants, and logistic and multinomial logistics regression analyses with interactions to determine whether and why any observed patterns in CRC screening behavior vary by race.

Status:

Completed

ELIGIBILITY:
Inclusion Criteria:

Study subjects must be a male or female veteran who has had one or more primary care visits at a VHA medical center in the past 2 years and is between the age of 50 and 75.

Exclusion Criteria:

Study subjects cannot be a VHA employee, deceased, have a colorectal cancer diagnosis, be enrolled in VA adult day care or nursing home, or have dementia.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care patients
Sampling Method: Probability Sample
Enrollment: 4644 (Actual)
Dates: Start 2006-03; Primary Completion 2007-05 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
colorectal cancer screening compliance | self-report or medical records documentation of either a fecal occult blood test (FOBT) in the past 15 months, a sigmoidoscopy or double contrast barium enema in the past 5.5 years, or a colonoscopy in the past 11 years

CONTACTS AND LOCATIONS:
Overall Officials: Melissa R. Partin, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Partin MR, Grill J, Noorbaloochi S, Powell AA, Burgess DJ, Vernon SW, Halek K, Griffin JM, van Ryn M, Fisher DA. Validation of self-reported colorectal cancer screening behavior from a mixed-mode survey of veterans. Cancer Epidemiol Biomarkers Prev. 2008 Apr;17(4):768-76. doi: 10.1158/1055-9965.EPI-07-0759. Epub 2008 Apr 1. PMID 18381474
- [Result] Burgess DJ, Powell AA, Griffin JM, Partin MR. Race and the validity of self-reported cancer screening behaviors: development of a conceptual model. Prev Med. 2009 Feb;48(2):99-107. doi: 10.1016/j.ypmed.2008.11.014. Epub 2008 Dec 11. PMID 19118570
- [Result] Partin MR, Burgess DJ, Halek K, Grill J, Vernon SW, Fisher DA, Griffin JM, Murdoch M. Randomized trial showed requesting medical records with a survey produced a more representative sample than requesting separately. J Clin Epidemiol. 2008 Oct;61(10):1028-35. doi: 10.1016/j.jclinepi.2007.11.015. Epub 2008 Jun 11. PMID 18550333
- [Result] Friedemann-Sanchez G, Griffin JM, Partin MR. Gender differences in colorectal cancer screening barriers and information needs. Health Expect. 2007 Jun;10(2):148-60. doi: 10.1111/j.1369-7625.2006.00430.x. PMID 17524008
- [Result] Burgess DJ, van Ryn M, Grill J, Noorbaloochi S, Griffin JM, Ricards J, Vernon SW, Fisher DA, Partin MR. Presence and correlates of racial disparities in adherence to colorectal cancer screening guidelines. J Gen Intern Med. 2011 Mar;26(3):251-8. doi: 10.1007/s11606-010-1575-7. Epub 2010 Nov 18. PMID 21088920
- [Result] Kodl MM, Powell AA, Noorbaloochi S, Grill JP, Bangerter AK, Partin MR. Mental health, frequency of healthcare visits, and colorectal cancer screening. Med Care. 2010 Oct;48(10):934-9. doi: 10.1097/MLR.0b013e3181e57901. PMID 20706162
- [Result] Partin MR, Noorbaloochi S, Grill J, Burgess DJ, van Ryn M, Fisher DA, Griffin JM, Powell AA, Halek K, Bangerter A, Vernon SW. The interrelationships between and contributions of background, cognitive, and environmental factors to colorectal cancer screening adherence. Cancer Causes Control. 2010 Sep;21(9):1357-68. doi: 10.1007/s10552-010-9563-0. Epub 2010 Apr 24. PMID 20419343
- [Result] Burgess DJ, Grill J, Noorbaloochi S, Griffin JM, Ricards J, van Ryn M, Partin MR. The effect of perceived racial discrimination on bodily pain among older African American men. Pain Med. 2009 Nov;10(8):1341-52. doi: 10.1111/j.1526-4637.2009.00742.x. PMID 20021596
- [Result] Powell AA, Burgess DJ, Vernon SW, Griffin JM, Grill JP, Noorbaloochi S, Partin MR. Colorectal cancer screening mode preferences among US veterans. Prev Med. 2009 Nov;49(5):442-8. doi: 10.1016/j.ypmed.2009.09.002. Epub 2009 Sep 8. PMID 19747502
- [Result] Griffin JM, Burgess D, Vernon SW, Friedemann-Sanchez G, Powell A, van Ryn M, Halek K, Noorbaloochi S, Grill J, Bloomfield H, Partin M. Are gender differences in colorectal cancer screening rates due to differences in self-reporting? Prev Med. 2009 Nov;49(5):436-41. doi: 10.1016/j.ypmed.2009.09.013. Epub 2009 Sep 16. PMID 19765609